CLINICAL TRIAL: NCT07223944
Title: A Phase 3 Safety and Efficacy Trial of FLT201 Gene Therapy in Patients With Gaucher Disease Type 1
Brief Title: A Gaucher Disease Gene Therapy Trial With FLT201
Acronym: GALILEO-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Spur Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLT201-03; 2025-520765-50-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Gaucher Disease Type 1
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FLT201 (Experimental): FLT201 is an advanced therapy investigational medicinal product (ATIMP) administered as a single intravenous infusion
  Interventions: Genetic: FLT201

INTERVENTIONS:
Genetic: FLT201 — FLT201 is a replication-incompetent single-stranded (ss) recombinant adeno-associated virus (AAV) vector. The vector is composed of a ss DNA genome packaged in an AAV-derived protein capsid.

SUMMARY:
This study is a Phase 3, non-randomized, multicenter, efficacy and safety study in adult patients with Gaucher disease Type 1, on stable treatment with enzyme replacement therapy (ERT) or substrate reduction therapy (SRT) for at least 2 years. The study aims to confirm the efficacy and safety of FLT201 in this population after discontinuation of ERT/SRT.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged ≥18 years at time of screening.
* Clinical diagnosis of Gaucher disease type 1
* Stable hemoglobin concentration at baseline
* Stable platelet count at baseline
* Receiving ERT or SRT without interruption for at least 2 years

Key Exclusion Criteria:

* Diagnosed or suspected Gaucher disease type 2 or type 3
* Positive for AAVS3 neutralizing antibodies.
* Abnormal lab values, conditions or diseases that would make the participant unsuitable for the study
* Positive pregnancy test or lactating
* History of hematopoietic stem cell transplant (HSCT)/bone marrow transplant or any solid organ transplant.
* History of receiving any gene therapy or cell therapy.
* History of total splenectomy. Note: Additional protocol defined Inclusion and Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of FLT201 | 1 Year
  Proportion of participants with stable hemoglobin concentration (decrease from baseline of no more than 1.5 g/dL) at Week 52